CLINICAL TRIAL: NCT00725192
Title: Sleep-directed Hypnosis As A Complement To CPT In Treating PTSD
Brief Title: Sleep-directed Hypnosis As A Complement To Cognitive Processing Therapy (CPT) In Treating Posttraumatic Stress Disorder (PTSD)
Acronym: Hypnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Trauma Recovery, St Louis (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Tara Galovski, University of Missouri- St. Louis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21AT004079-01A1 (NIH)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Posttraumatic Stress Disorder; Physical Assault; Physical Abuse; Sexual Assault; Sexual Abuse; Interpersonal Assault; Cognitive Processing Therapy; Sleep Impairment; Insomnia; Hypnosis
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cognitive Processing Therapy
  Interventions: Behavioral: Cognitive Processing Therapy
- 2 (Experimental): Hypnosis plus Cognitive Processing Therapy.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Clients will receive between 12 sessions of Cognitive Processing Therapy.
Behavioral: Hypnosis — PArticipants will receive 3 sessions of hypnosis to specifically target sleep impairment.
  Arms: 2

SUMMARY:
Sleep impairment is the most often reported of the 17 PTSD symptoms and is considered one of the most refractory to treatment. This study proposes the use of sleep-directed hypnotherapy to address sleep issues as a complementary element to empirically supported Cognitive Processing Therapy (CPT) in treating PTSD in sexual and physical assault survivors. Specifically the study aims to: 1) compare the results of sleep-directed hypnosis plus CPT with CPT only, 2) to assess the relationship between sleep and PTSD symptoms, 3) to examine relationships between sleep improvement, PTSD symptom improvement, and the therapeutic elements (hypnosis, exposure, cognitive therapy) to determine mechanisms of action in the intervention, 4) to assess the relationship between sleep and physical reactivity to trauma-related cues and to other stimuli.

DETAILED DESCRIPTION:
Cognitive Processing Therapy (CPT) has demonstrated significant empirical support in treating victims of sexual assault suffering from Posttraumatic Stress Disorder (PTSD) throughout its program of research at the University of Missouri - St. Louis. Similarly to the larger treatment outcome literature, these clinical trials have revealed a portion of participants whose sleep remains refractory to treatment even after conclusion of a full course of treatment.

In fact, the specific causes of sleep disturbance in posttraumatic stress disorder (PTSD) sufferers, the most prominent of which are insomnia and nightmares, have not been determined. However, sleep impairment is the most often reported of the 17 PTSD symptoms and is considered one of the most refractory to treatment. It is theorized that PTSD sleep impairment relates to the hypervigilance inherent in PTSD such that sleep is disrupted by the perception that vigilance (in response to perceived threat) must be maintained at night. Sleep impairment seen in PTSD sufferers may then result from increased physiological arousal associated with chronic hypervigilance. Hypnosis provides deep relaxation which is hypothesized to decrease overall hyperarousal. Nightmares and trauma cues can further disrupt sleep through learning and conditioning. PTSD sufferers may learn to associate nighttime cues with danger and conditioned emotional responses to these cues may disrupt sleep. Detecting relatively innocuous environmental stimuli (i.e. normal nighttime noises) while trying to fall asleep and interpreting them as dangerous increases arousal. Hyperarousal interferes with sleep and has been identified as causal in the development of non-PTSD insomnia. Beyond decreases in general hyperarousal, an additive benefit of the hypnotic trance and the use of post-hypnotic suggestion would be the facilitation of new learning such that bedroom stimuli could become associated with pleasant, restful images. The use of hypnosis as a complement to CPT, an empirically supported, cognitive-behavioral intervention developed to treat PTSD, could specifically remediate 1.) sleep onset and maintenance deficits, 2) the frequency and intensity of parasomnia episodes, and 3.) cumulative sleep deprivation. Acquisition of the skill of self-hypnosis will provide PTSD sufferers with a tool to regain normal and restorative sleep patterns. Restoring sleep will enhance the efficacy of CPT in remediating psychiatric symptoms (PTSD and major depression), reduce overall physiological reactivity, increase psychosocial functioning, and decrease somatization.

This study proposes the use of sleep-directed hypnotherapy as a complementary element to the empirically supported CPT in treating PTSD in sexual and physical assault survivors. Specifically:

Aim 1: Compare the results of sleep-directed hypnosis + CPT (hypCPT) versus CPT-only (CPT) within a sample of female sexual/physical assault survivors. It is hypothesized that the hypCPT group will show significantly greater improvement on overall PTSD severity, concurrent psychopathology, and overall sleep impairment.

Aim 2: Assess the relationship between sleep and PTSD sxs. Specifically, identify temporal and directional relationships between elevations in PTSD symptoms and increases in sleep impairment while accounting for daily life stressors.

Aim 3: Evaluate improvements with respect to the process of therapy. Specifically, examine relationships between sleep improvement, PTSD symptom improvement, and the therapeutic elements (hypnosis, exposure, cognitive therapy) to determine mechanisms of action in the intervention. It is specifically hypothesized that improvements in sleep will be positively and temporally related to improvements in PTSD symptomatology throughout treatment. Further, overall decreases in sleep impairment will indicate a temporal, positive relationship to overall improvements in psychosocial functioning and health-related concerns.

Aim 4: Assess the relationship between sleep and psychophysiological reactivity to trauma-related cues and to an auditory startle probe. It is hypothesized that impairment in sleep onset and maintenance, frequency/intensity of parasomnia episodes, and overall sleep deprivation will be positively related to elevations in psychophysiological reactivity (heart-rate, skin conductance, and facial EMG) during a scripted-imagery paradigm and an auditory startle paradigm. It is further hypothesized that decreases in sleep impairment will be positively related to decreases in physiological reactivity across hypCPT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be at least three months post-crime at the time of their participation and will have been diagnosed with PTSD. Participants will score at least a "3" on the CAPS symptom of sleep impairment. This score is indicative of clinically significant symptomatology on any PTSD symptom. There is no upper limit on time since the trauma for participation.

Exclusion Criteria:

* Exclusion criteria for participants include psychosis, mental retardation, active suicidality, parasuicidality, or current addiction to drugs or alcohol. In the case of apparent illiteracy, we will try to accommodate the individual as much as possible to maximize success in the program. In addition, participants cannot be in a currently abusive relationship or being stalked. For marital rape or domestic violence, the participant must have been out of the relationship for at least three months. Participants can have received any therapy in the past with the exception of CPT. They may be receiving concurrent therapy as long as it is not trauma-focused. Allowing subjects to continue with concurrent therapy offers them the option to continue with established supports and more closely mimics clinical practice and the generalizability of the results. Participants will be asked to monitor and adhere to several behaviors that significantly impact sleep and may introduce error into the study aims. Inability or unwillingness to comply the the following will constitute exclusion criteria: Participants will be asked not to increase sleep medications, but to continue usual practice. This usage will be monitored on a daily basis on the sleep diaries. Daytime sleeping or naps will be monitored on the daily diaries and used as an outcome measure as naps are utilized less and less frequently across time in a number of insomnia treatment studies. Participants will also be asked to keep alcohol consumption to no more than 14 servings per week with no more than 5 servings on any given day. We will also ask participants to consume no more than 500 mg of caffeine on a daily basis and to refrain from caffeine consumption after 6 pm. We will further ask participants to maintain their bedtime and rise time during the work week and to not vary these times by more than one hour on days off. Participants will record bedtime and rise time on their daily diaries. Participants will be asked to maintain these sleep-related behaviors for the duration of therapy - approximately 8-10 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Good end-state functioning: Beck Depression Inventory-II and Posttraumatic Distress Scale Scores | 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tara Galovski, PhD, Principal Investigator — Center for Trauma Recovery, University of Missouri- St. Louis
Locations (1):
- Center for Trauma Recovery, St Louis, Missouri, United States

REFERENCES:
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Alpert E, Carpenter JK, Smith BN, Woolley MG, Raterman C, Farmer CC, Kehle-Forbes SM, Galovski TE. Leveraging observational data to identify in-session patient and therapist predictors of cognitive processing therapy response and completion. J Trauma Stress. 2023 Apr;36(2):397-408. doi: 10.1002/jts.22924. Epub 2023 Mar 29. PMID 36987703